CLINICAL TRIAL: NCT03434262
Title: Molecularly-Driven Doublet Therapy for All Children With Refractory or Recurrent CNS Malignant Neoplasms and Young Adults With Refractory or Recurrent SHH Medulloblastoma
Brief Title: SJDAWN: St. Jude Children's Research Hospital Phase 1 Study Evaluating Molecularly-Driven Doublet Therapies for Children and Young Adults With Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJDAWN; NCI-2018-00284 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Ependymoma; Anaplastic Ganglioglioma; Anaplastic Meningioma; Anaplastic Oligodendroglioma; Pleomorphic Xanthoastrocytoma, Anaplastic; Atypical Teratoid/Rhabdoid Tumor; Brain Cancer; Brain Tumor; Central Nervous System Neoplasms; Choroid Plexus Carcinoma; CNS Embryonal Tumor With Rhabdoid Features; Ganglioneuroblastoma of Central Nervous System; CNS Tumor; Embryonal Tumor of CNS; Ependymoma; Glioblastoma; Glioma; Glioma, Malignant; Medulloblastoma; Medulloblastoma; Unspecified Site; Medulloepithelioma; Neuroepithelial Tumor; Neoplasms; Neoplasms, Neuroepithelial; Papillary Tumor of the Pineal Region (High-grade Only); Pediatric Brain Tumor; Pineal Parenchymal Tumor of Intermediate Differentiation (High-grade Only); Pineoblastoma; Primitive Neuroectodermal Tumor; Recurrent Medulloblastoma; Refractory Brain Tumor; Neuroblastoma. CNS; Glioblastoma, IDH-mutant; Glioblastoma, IDH-wildtype; Medulloblastoma, Group 3; Medulloblastoma, Group 4; Glioma, High Grade; Neuroepithelial Tumor, High Grade; Medulloblastoma, SHH-activated and TP53 Mutant; Medulloblastoma, SHH-activated and TP53 Wildtype; Medulloblastoma, Chromosome 9q Loss; Medulloblastoma, Non-WNT Non-SHH, NOS; Medulloblastoma, Non-WNT/Non-SHH; Medulloblastoma, PTCH1 Mutation; Medulloblastoma, WNT-activated; Ependymoma, Recurrent; Glioma, Recurrent High Grade; Glioma, Recurrent Malignant; Embryonal Tumor, NOS; Glioma, Diffuse Midline, H3K27M-mutant; Embryonal Tumor With Multilayered Rosettes (ETMR); Ependymoma, NOS, WHO Grade III; Ependymoma, NOS, WHO Grade II; Medulloblastoma, G3/G4; Ependymoma, RELA Fusion Positive
Keywords: ATRT; Brain Tumors in Adolescents; Brain Tumors in Children; Brain Tumors in Young Adults; CDK4 amplification; CDK 4/6; CDK 4/6 inhibitor; CDK 4/6 pathway; CDK 4/6/cyclin/RB/E2F pathway; CDK6 amplification; CyclinD1; DAWN; D-type Cyclins; Hedgehog pathway inhibitor; HGG; MAPK pathway; MEK; MEK inhibitor; MEK1; MEK2; Mekinist; Molecular; Molecular therapy; MYC amplification; PTCH1; Rare brain tumor; Recurrent ATRT; Recurrent brain tumor; Recurrent ependymoma; Recurrent high grade glioma; Recurrent malignant glioma; Recurrent medulloblastoma; Refractory brain tumor; Small molecule inhibitor; SMO antagonist; Smoothened protein; Sonic hedgehog; Combination therapy
MeSH Terms: conditions — Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Rhabdoid Tumor; Brain Neoplasms; Central Nervous System Neoplasms; Choroid Plexus Carcinoma; Glioblastoma; Glioma; Medulloblastoma; Neuroectodermal Tumors, Primitive; Neoplasms, Neuroepithelial; Neoplasms; Pinealoma; Pyloric Stenosis, Hypertrophic; Recurrence; Neoplasms, Germ Cell and Embryonal; Lymphoma, Follicular; Microphthalmia, Isolated, with Coloboma 5 | interventions — Gemcitabine; ribociclib; sonidegib; trametinib; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This is a phase 1 limited dose escalation to define RP2D of the doublets with an early expansion cohort to evaluate preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: ribociclib + gemcitabine (Experimental): Stratum A participants with a diagnosis of refractory or recurrent medulloblastoma (Group 3/4) or refractory or recurrent ependymoma. (including: ependymoma, not otherwise specified (NOS), WHO Grade III; ependymoma, RELA fusion positive; anaplastic ependymoma; ependymoma, NOS, WHO grade II). They receive combination treatment with ribociclib and gemcitabine. They may also receive growth therapy support with filgrastim.
  Stratum A has completed all the necessary accrual
  Interventions: Drug: Gemcitabine; Drug: ribociclib; Biological: filgrastim
- B: ribociclib + trametinib (Experimental): Stratum B participants with a diagnosis of one of the following refractory or recurrent CNS diseases: medulloblastoma, [sonic hedgehog (SHH)- or WNT-activated];; high grade glioma (including: high grade glioma, (NOS), WHO Grade III or IV; anaplastic astrocytoma, IDH mutant; glioblastoma, IDH-wildtype; glioblastoma, IDH-mutant; diffuse midline glioma, H3K27-mutant; anaplastic oligodendroglioma, IDH mutant and 1p/19q-codeleted; anaplastic pleomorphic xanthoastrocytoma); select CNS embryonal tumors (including: embryonal tumors with multilayered rosettes, C19MC-altered; embryonal tumors with multilayered rosettes, NOS; medulloepithelioma; CNS neuroblastoma; CNS ganglioneuroblastoma; CNS embryonal tumor, NOS; atypical teratoid/rhabdoid tumor; CNS embryonal tumor with rhabdoid features). They receive combination treatment with ribociclib and trametinib.
  Stratum B has completed all the necessary accrual
  Interventions: Drug: ribociclib; Drug: trametinib
- C: ribociclib + sonidegib (Experimental): Stratum C participants with refractory or recurrent medulloblastoma (SHH-activated) >6 months off smoothened inhibitor, presence of 9q loss or PTCH1 mutant, skeletally mature. They received combination treatment with ribociclib and sonidegib.
  Stratum C is being closed due to low accrual
  Interventions: Drug: ribociclib; Drug: sonidegib

INTERVENTIONS:
Drug: Gemcitabine — Given intravenously (IV).
  Other Names: Gemzar®
  Arms: A: ribociclib + gemcitabine
Drug: ribociclib — Given orally (PO).
  Other Names: LEE011; LEE-011; KISQALI®
Drug: sonidegib — Given PO.
  Other Names: LDE225; LDE-225; ODOMZO®
  Arms: C: ribociclib + sonidegib
Drug: trametinib — Given PO.
  Other Names: TMT212; TMT-212; MEKINIST(TM)
  Arms: B: ribociclib + trametinib
Biological: filgrastim — Given subcutaneously (SQ).
  Other Names: G-CSF
  Arms: A: ribociclib + gemcitabine

SUMMARY:
Approximately 90% of children with malignant brain tumors that have recurred or relapsed after receiving conventional therapy will die of disease. Despite this terrible and frustrating outcome, continued treatment of this population remains fundamental to improving cure rates. Studying this relapsed population will help unearth clues to why conventional therapy fails and how cancers continue to resist modern advances. Moreover, improvements in the treatment of this relapsed population will lead to improvements in upfront therapy and reduce the chance of relapse for all. Novel therapy and, more importantly, novel approaches are sorely needed. This trial proposes a new approach that evaluates rational combination therapies of novel agents based on tumor type and molecular characteristics of these diseases. The investigators hypothesize that the use of two predictably active drugs (a doublet) will increase the chance of clinical efficacy. The purpose of this trial is to perform a limited dose escalation study of multiple doublets to evaluate the safety and tolerability of these combinations followed by a small expansion cohort to detect preliminary efficacy. In addition, a more extensive and robust molecular analysis of all the participant samples will be performed as part of the trial such that we can refine the molecular classification and better inform on potential response to therapy. In this manner the tolerability of combinations can be evaluated on a small but relevant population and the chance of detecting antitumor activity is potentially increased. Furthermore, the goal of the complementary molecular characterization will be to eventually match the therapy with better predictive biomarkers.

PRIMARY OBJECTIVES:

* To determine the safety and tolerability and estimate the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) of combination treatment by stratum.
* To characterize the pharmacokinetics of combination treatment by stratum.

SECONDARY OBJECTIVE:

* To estimate the rate and duration of objective response and progression free survival (PFS) by stratum.

DETAILED DESCRIPTION:
Patients will be stratified by the molecular and histologic characteristics of their tumor to one of three treatment strata.

STRATUM A:

* Combination Treatment: ribociclib and gemcitabine.
* Patient Population: Participants with a diagnosis of refractory or recurrent medulloblastoma (Group 3/4) or refractory or recurrent ependymoma (including: ependymoma, not otherwise specified (NOS), WHO Grade III; ependymoma, RELA fusion positive; anaplastic ependymoma; ependymoma, NOS, WHO grade II).

STRATUM B:

* Combination Treatment: ribociclib and trametinib.
* Patient Population: Participants with a diagnosis of one of the following refractory or recurrent CNS diseases: medulloblastoma [sonic hedgehog (SHH)], medulloblastoma (WNT), high grade glioma (including: high grade glioma, (NOS), WHO Grade III or IV; anaplastic astrocytoma, IDH mutant; glioblastoma, IDH-wildtype; glioblastoma, IDH-mutant; diffuse midline glioma, H3K27-mutant; anaplastic oligodendroglioma, IDH mutant and 1p/19q-codeleted; anaplastic pleomorphic xanthoastrocytoma) or select central nervous system (CNS) embryonal tumors (including: embryonal tumors with multilayered rosettes, C19MC-altered; embryonal tumors with multilayered rosettes, not otherwise specified (NOS); medulloepithelioma; CNS neuroblastoma; CNS ganglioneuroblastoma; CNS embryonal tumor, NOS; atypical teratoid/rhabdoid tumor; CNS embryonal tumor with rhabdoid features).

STRATUM C:

* Combination Treatment: ribociclib and sonidegib.
* Patient Populations: Participants with refractory or recurrent medulloblastoma (SHH) >6 months off smoothened inhibitor, presence of 9q loss or PTCH1 mutant, skeletally mature.

The rolling 6 design will be used separately in each stratum to estimate the MTD or RP2D and determine the dose-limiting toxicity (DLT) of the combination of escalating doses. Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity. Stratum A participants may continue therapy past 24 months in absence of disease progression or unacceptable toxicity.

Patients will receive doublet therapy in cycles of 28 days. The dose-limiting toxicity (DLT)-evaluation period will consist of the first cycle (i.e. first 4 weeks of therapy). Research participants will be evaluated at least once a week during the DLT-evaluation period and at regular intervals thereafter. Standard (e.g., physical exam, blood tests, and disease evaluations) tests will be obtained at regular intervals. Research-associated evaluations (e.g., pharmacokinetic studies, etc.) will also be obtained during therapy. Treatment may be continued for up to 2 years in the absence of disease progression or unacceptable toxicity. Stratum A participants may continue past 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Potential participants will first be screened using the screening inclusion/exclusion shown below. If they meet the requirements of the screening phase, they will then be evaluated for enrollment based on the overall study's inclusion criteria as well as the stratum-specific inclusion/exclusion criteria for the applicable stratum, all of which are shown below.

SCREENING INCLUSION CRITERIA - ALL PARTICIPANTS:

* Participants with recurrent, progressive, or refractory brain tumors.
* Age ≥ 1 year and < 25 years at the time of screening. Exception: Participants with recurrent, progressive, or refractory Medulloblastoma and are ≥ 1 and < 40 years of age at the time of study screening are eligible for screening.
* Participants and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

SCREENING EXCLUSION CRITERIA - ALL PARTICIPANTS:

* Participants with a diagnosis of recurrent, progressive, or refractory low grade glioma (LGG).
* Previous exposure to a CDK4/6 inhibitor (palbociclib, abemaciclib, or ribociclib).
* Participants with a history of clinically significant, uncontrolled heart disease and/or repolarization abnormalities.
* Participants with any history of QTc prolongation (i.e. QTc interval of > 450 msec).

Participants who meet the requirements of the screening phase will then be evaluated for enrollment based on the overall study's inclusion criteria as well as the stratum-specific inclusion/exclusion criteria for the applicable stratum, all of which are shown below.

INCLUSION CRITERIA - OVERALL STUDY - ALL PARTICIPANTS:

* Evaluable disease, as defined as meeting any of the following:

  * Patients who have measurable disease
  * Patients with radiologically discernible but non-measurable lesions (i.e. leptomeningeal disease)
  * Patients with CSF positive disease
* Participants must have received their last dose of anticancer therapy (including experimental) at least 4 weeks prior to study enrollment.

  * Note: Participants must have relapsed with recurrent, progressive or refractory disease on or after any prior anticancer therapy.
* Participants must have had their last fraction of radiation at least 4 weeks prior to study enrollment. Participants who received radiation therapy for palliation must have had their last fraction of radiation at least 2 weeks prior to study enrollment.

  * Note: Participants must have relapsed with recurrent, progressive or refractory disease after any prior radiation therapy that is not considered palliative. Palliative radiation therapy is defined as local small port RT to alleviate and/or palliate symptoms. (CSI, whole brain RT, large field/port RT, or large field/port multilevel spinal RT will not be considered palliative at any dose.)
* Participants who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to study enrollment with no plans for escalation.
* Participants who are receiving known strong inducers and/or strong inhibitors of CYP3A4/5, drugs that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5, and medications that carry a known risk for QT prolongation must discontinue these drugs at least 7 days prior to study enrollment.
* Participants must discontinue herbal preparations, herbal medication, and dietary supplements, with the exception of multivitamins, at least 7 days prior to study enrollment.
* Participants must be able to swallow medication. It is acceptable to administer medication via a g-tube if participant has a g-tube. It is not acceptable to place a g-tube for the purpose of delivering study medication.
* Participants must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of at least 50 and, in the opinion of the investigator, a minimum life expectancy of at least 6 weeks at the time of study enrollment.

  * Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participant must have adequate bone marrow and organ function defined as:

  * ANC ≥ 1000/mm3 without growth factor support within 7 days of the test
  * Platelet count ≥ 50,000/mm^3 without support of a platelet transfusion within 7 days of the test
  * Hemoglobin ≥ 8.0 g/dL without support of a blood transfusion within 7 days of the test
  * Creatinine clearance ≥ 70 mL/min/1.73 m^2 or serum creatinine ≤ the maximum serum creatinine based on age/gender (threshold creatinine values derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention or creatinine clearance ≥70 mL/min/1.73 m^2).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN. For the purposes of eligibility the ULN of ALT and AST is 45 U/L.
  * Total bilirubin ≤ ULN or if > ULN then direct bilirubin ≤ 1.5xULN.
* Participants and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

EXCLUSION CRITERIA - OVERALL STUDY - ALL PARTICIPANTS:

* Participants receiving any other investigational agents.
* Participants with other clinically significant medical disorders (serious infections or significant cardiac, pulmonary, hepatic, psychiatric, GI disease, or other organ dysfunction) that in the investigator's judgment could compromise their ability to tolerate or absorb protocol therapy or would interfere with the study procedures or results.
* Female participants who are breastfeeding a child.
* Participants with QTc interval of > 450 msec on screening ECG.
* Participants with a pathogenic somatic or known germline retinoblastoma (RB1) gene mutation.

(A) INCLUSION CRITERIA - STRATUM A PARTICIPANTS ONLY:

* Participants with recurrent, progressive, or refractory Non-WNT Non-SHH (NWNS) Medulloblastoma or Ependymoma as confirmed through central pathology review.
* Age ≥ 1 year and < 25 years at the time of enrollment.
* Female participants of childbearing potential must have a negative pregnancy test at the time of enrollment on this study and be willing to use a highly effective method of contraception throughout the study and for 16 weeks after discontinuation of the study drug.
* Male participants of child fathering potential must be willing to use medically acceptable form of contraception during treatment and for 16 weeks after stopping treatment.

(A) EXCLUSION CRITERIA - STRATUM A PARTICIPANTS ONLY:

* Participants with subependymoma or myxopapillary ependymoma.

(B) INCLUSION CRITERIA - STRATUM B PARTICIPANTS ONLY:

* Participants with recurrent, progressive, or refractory CNS tumors as confirmed through central pathology review and whose diagnosis is being treated on this study.
* Age ≥ 1 year and < 25 years at the time of study enrollment.
* Must meet the following weight and BSA restrictions:

  * For enrollment on dose levels 0A, must have a weight ≥16kg and <32kg.
  * For enrollment on dose level 0B, must have a weight of ≥32kg and BSA ≥ 0.55m^2.
  * For enrollment on dose level 1, must have a weight ≥16kg and BSA ≥0.55m^2.
  * For enrollment on dose level 2, must have a weight ≥16kg and BSA≥ 0.63m^2
  * For enrollment on dose levels 3 or 4A, must have a weight ≥16kg
  * For enrollment on dose levels 4B or 5, must have a weight ≥20kg and ≤106kg
* Participant must be able to swallow trametinib tablets.
* Female participants of childbearing potential must have a negative pregnancy test at the time of enrollment on this study and be willing to use a highly effective method of contraception throughout the study and for 16 weeks after discontinuation of the study drug.
* Male participants of child fathering potential must be willing to use medically acceptable form of contraception during treatment and for 16 weeks after stopping treatment.

(B) EXCLUSION CRITERIA - STRATUM B PARTICIPANTS ONLY: Participants eligible for this study must NOT meet ANY of the following criteria.

* Participants with Low Grade Glioma (LGG) or Diffuse Intrinsic Pontine Glioma (DIPG).
* Previous exposure to a MEK inhibitor (i.e. trametinib, selumetinib).
* Participants with abnormal LVEF on screening, defined as > 10% below lower limit of normal on screening.
* Participants with retinal vein occlusion (RVO).
* Previous exposure to a MEK inhibitor (i.e., trametinib, selumetinib.

(C) INCLUSION CRITERIA - STRATUM C PARTICIPANTS ONLY:

* Participants with recurrent, progressive, or refractory SHH Medulloblastoma and presence of either a or b as confirmed by central pathology review of the tumor specimen: a) copy number loss of 9q b) PTCH1 mutation and whose diagnosis is being treated on this study.
* Age ≥ 10 years and <40 years at the time of study enrollment.
* Participant must be skeletally mature as defined as females with a bone age ≥ 15 years (180 months) and males with a bone age ≥ 17 years (204 months). This includes participants that are within 2 standard deviations of this value (i.e. if SD = 11 months on bone age; then a male patient who has a bone age of 182 months would be eligible; or a female patient with a bone age of 158 months.)
* Female participants of childbearing potential must have a negative pregnancy test at the time of enrollment on this study and be willing to use a highly effective method of contraception throughout the study and for 8 months after discontinuation of the study drug.
* Male participants of child fathering potential must be willing to use medically acceptable form of contraception during treatment and for 8 months after stopping treatment.

(C) EXCLUSION CRITERIA - STRATUM C:

* Exposure to smoothened inhibitor (vismodegib, sonidegib) within the last 6 months.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Estimate the Maximum tolerated dose (MTD)/Recommended Phase 2 Dose (RP2D) of each doublet by stratum | 1 month after start of therapy
  The MTD is empirically defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. The MTD estimate will not be available, if the lowest dose level studied is too toxic or the highest dose level studied is considered safe. In the latter case, the highest studied safe dose will be considered the recommended phase 2 dose (RP2D). The MTD estimation will be limited to evaluable patients and toxicity assessments from course 1 (28 days).
Pharmacokinetics of combination treatment: Stratum A | Course 1: Days -1, 0, 1 and 15 and 16; Course 2: Day 1
  Plasma concentration will be provided.
Pharmacokinetics of combination treatment: Stratum B | Course 1: Days 1, 2, 3, 14 and 15
  Plasma concentration will be provided.
Pharmacokinetics of combination treatment: Stratum C | Course 1: Days -1, 0, 1, 2, 21, 22 and 28; Course 2: Day 1
  Plasma concentration will be provided.

SECONDARY OUTCOMES:
Response rate by stratum | Up to 1 year after completion of therapy (up to 3 years after start of therapy)
  The response rate, defined as the rate of complete response (CR) or partial response (PR), and long-term stable disease (SD) will be calculated as the percentage of confirmed responders among all response assessable patients. These rates as well as their exact confidence intervals will be provided and will be summarized by each response category (i.e., CR, PR, and SD). Descriptive summaries of response per dose level may also be provided. Subjects without an assessment will be considered non-responders.
Duration of objective response by stratum | Up to 1 year after completion of therapy (up to 3 years after start of therapy)
  Duration of response defined as the time from the initial documented response (CR or PR) to the first confirmed progressive disease (PD). We will use progression free survival (PFS) for describing duration of SD. Subjects without a documented progression will be censored at the time of their last tumor assessment. Duration of Response will be assessed using the Kaplan-Meier method to calculate the median time as well as the proportion remaining progression free at given time points. The corresponding 95% confidence intervals will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Giles W. Robinson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — https://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042a579a1474aa7f29de3b5=2